CLINICAL TRIAL: NCT00097656
Title: MOTOR: Maternal Oral Therapy to Reduce Obstetric Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NIDCR-14577; U01DE014577 (NIH); 5U01DE014577 (NIH)
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Pregnancy Related; Periodontitis; Premature Birth
MeSH Terms: conditions — Periodontitis; Premature Birth | interventions — Random Allocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Periodontal Treatment (Experimental): maternal periodontal therapy
  Interventions: Other: multi-center, randomized, controled periodontal therapy

INTERVENTIONS:
Other: multi-center, randomized, controled periodontal therapy — periodontal therapy
  Other Names: Periodontal Therapy

SUMMARY:
The purpose of this study is to determine whether maternal periodontal therapy (tooth cleaning) decreases the rate of preterm deliveries at <37 weeks gestation and to determine the effects of maternal periodontal therapy on the birth weight of infants born less than 37 weeks gestation.

DETAILED DESCRIPTION:
STUDY DESIGN:

The intervention is designed as a multi-center, randomized, controlled, clinical trial to determine the effects of periodontal therapy on the rate of preterm birth. Study participants will be assigned to one of two study arms. All pregnant women who present to the designated Obstetrical (OB) clinics are potential subjects for this study. A total of 1800 patients will be enrolled at 3 performance sites, enrolling about 600 subjects at each site at a rate of about 171 subjects/year at each site, randomly assigning these subjects to one of 2 treatment arms. Randomization will be performed using a computer-generated assignment scheme designed and performed in a masked manner by the data coordinating center. Each performance site will enroll about 300 subjects into each treatment group using the intent-to-treat principle, obtaining follow-up on all subjects. In treatment Group 1 participants will be assigned to standard localized periodontal therapy of scaling and root planning with subgingival polishing between three and six months of gestation. Group 2 will receive the same local periodontal therapy immediately following delivery.

MASKING:

The dental examiner will not be aware of the randomization treatment assignments of participants until after a complete baseline periodontal examination has been conducted. The study protocol allows the dental examiner to know the treatment assignment of participants but this knowledge will not affect the assessment of the primary obstetric outcome of the study. OB personnel or individuals collecting OB data will be masked as to dental treatments. At delivery the second dental exam will be made without the examiner knowing the pregnancy outcome.

PRIMARY/SECONDARY OUTCOME MEASURES:

The primary outcome is preterm delivery at less than 37 weeks gestational age, as determined by ultrasound dating. Secondary outcomes include (1) preterm delivery less than 35 weeks, (2) weight for gestational age, and (3) neonatal morbidity/mortality. It is our central hypothesis that mothers with periodontitis that receive periodontal treatment during the second trimester of pregnancy will experience a lower rate of preterm delivery at <37 weeks and secondarily <35 weeks; that periodontal treatment of these pregnant mothers will result in an increase in the weight for gestational age of deliveries occurring less than 37 weeks gestational age and reduce neonatal morbidity and mortality. We will determine the effects of periodontal therapy on the rate of preterm birth at GA<37 weeks as the principal outcome and on mean birth weight among neonates with GA<35 weeks, as a secondary outcome adjusting for race, gender and gestational age.

POTENTIAL CONFOUNDERS AND COVARIATES:

There are many potential risk factors that relate to preterm birth and growth restriction that need to be considered in this investigation. There are also exposures, effect modifiers and covariates that influence periodontal disease status and preterm birth. Data will be collected on the major variables of interest to include race, age, smoking, previous preterm delivery, first births, bacterial vaginosis, chorioamnionitis, sexually transmitted diseases (STDs), antibiotic usage, socioeconomic status (SES) and substance abuse. In addition we will measure fetal fibronectin and collect vaginal smears to examine for potential subclinical vaginosis. Detailed information will be collected on these potential factors and used to assure that randomization has effectively balanced risk between treatment arms and to permit post-hoc assessments.

PLAN FOR MONITORING:

There will be an administrative Steering committee consisting of the Obstetric and Periodontal Principal Investigator(PI) from each clinical site, the NIDCR co-investigators and the Data and Statistical Coordinating Center (DSCC) investigators. The Steering committee will meet twice the first year and once a year thereafter. Study coordinators will also attend one of the two annual meetings. Data will be collected on dental, obstetric and neonatal outcomes by the data & statistical coordinating center, monitoring weekly for adverse events. The DSCC will be collating adverse events and safety data centrally to provide safety assessment reports to the DSMB. The DSMB will monitor outcomes and adverse events and assure maternal and infant safety and provide feedback to NIDCR every 6 months or as needed.

ADVERSE EVENTS:

The dental examiner will conduct a comprehensive oral soft tissue (cancer screening) and periodontal examination at baseline and at post partum. Following enrollment mothers will be followed up by, OB surveillance through parturition, a post-delivery dental follow-up and neonatal surveillance that includes chart review after discharge. All of these provide an opportunity to detect and monitor adverse events. All reported and observed serious adverse events will be documented on an adverse event case report form describing the onset, duration, severity, assessment of causality and relationship to treatment intervention. This will be followed until resolution. A member of the investigative team will review subject's OB charts on a weekly basis to note any adverse events or treatment provided (outside of routine). In addition all neonatal discharge summary findings will be collected to monitor any adverse neonatal morbidity such as neonatal sepsis and necrotizing enterocolitis. Any dental treatment will be noted in the subject's clinical record to be reviewed by the dental examiner.

PLAN FOR DATA ANALYSIS:

The details of the analysis plan appear in the body of the protocol, and are summarized here. The incidence of preterm birth as the principal outcome will be evaluated using a chi-square test. Approximately 240 cases are expected at gestational age (GA)<35 weeks. Success of randomization for possible confounders will be evaluated by logistic regression models. Significance will be indicated by an alpha level of 0.05. Mean birth weight among preterm babies will be analyzed for correlations and significant differences between study arms using a non-parametric test (Kruskal-Wallis test) Parametric (regression) models will be used to adjust for gestational age and other factors.]. Analyses will be conducted using the intent to treat philosophy. Data will be collected on a series of potential risk factors, covariates, confounders and effect modifiers that may influence the primary and secondary outcomes or periodontal status. Any unbalanced distribution of risks or exposures will be included in the regression model analysis. Adverse event data will be reported regularly. Interim analyses for efficacy will be conducted after 600 and 1200 completed pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Willing to be randomized and complete treatment protocols and provide informed consent
* Planning on prenatal care and delivery at the enrollment center
* Pregnant and able to complete periodontal treatment prior to 236 weeks gestation
* At least 16 years old at enrollment
* Minimum of 20 teeth present
* Three (3) or more periodontal sites with > 3mm clinical attachment loss

Exclusion Criteria:

* Multiple gestation
* Positive history of HIV infection, AIDS, autoimmune disease, or diabetes (gestational diabetes is acceptable)
* Any medical contraindication to periodontal probing or periodontal treatment that would require antibiotic prophylaxis, (e.g., congenital heart disease, use of Phen- fen for weight loss without a clear

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2004-02; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Birth at less than 37 weeks gestational age | 37 weeks gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Steven Offenbacher, DDS PhD MMS, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Offenbacher S, Beck JD, Jared HL, Mauriello SM, Mendoza LC, Couper DJ, Stewart DD, Murtha AP, Cochran DL, Dudley DJ, Reddy MS, Geurs NC, Hauth JC; Maternal Oral Therapy to Reduce Obstetric Risk (MOTOR) Investigators. Effects of periodontal therapy on rate of preterm delivery: a randomized controlled trial. Obstet Gynecol. 2009 Sep;114(3):551-559. doi: 10.1097/AOG.0b013e3181b1341f. PMID 19701034